CLINICAL TRIAL: NCT02274350
Title: The Herlev Hospital Post Radiation Therapy for Localized Prostate Cancer Database for Sexual Side Effects
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anders Frey, research assistant, Herlev Hospital
Other Study IDs: HEH-2014-091
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Cancer of the Prostate
Keywords: prostate cancer; radiation therapy; sexual side effects
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- radiation therapy: Patients treated with either external beam radiation therapy or brachie therapy for localized prostate cancer
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Radiation therapy either in the form of external beam radiation or radioactive gold seeds planted directly in the prostate.

SUMMARY:
The aim of this study is:

* To investigate which sexual side effects occur after external beam radiation therapy and brachie therapy
* To investigate how many patients are affected
* To investigate if there is a time dependency for the severity of the sexual side effects
* To investigate if there is a dose dependency for the severity of the sexual side effects
* To find predicting and associated factors for the discovered sexual side effects to help identifying patients at risk

DETAILED DESCRIPTION:
Aim:

According to the European Association of Urology guidelines radical prostatectomy (RP) and external beam radiation therapy (EBRT) are considered equal treatments with curative intends, for localized prostate cancer [1]. Another type of radiation therapy used to treat localized prostate cancer is brachytherapy (BT). After both RP and EBRT some patients suffer a degree of erectile dysfunction (ED) and urinary incontinence (UI) [2-5]. However, current evidence shows that rates are lower with EBRT [4,5]. Unfortunately, EBRT hold the potential for late-onset toxicity and can, in a small percentage of the patients, lead to secondary genitourinary or gastrointestinal cancers [5]. In a recent study of RP patients at Herlev hospital, the investigators found that many patients, in addition to ED and UI, also suffered from UI during sexual activity, Orgasmic dysfunction, and penile morphological and sensory changes [6]. Only few studies have investigated these side effects in EBRT and BT patients.

The aim for this study is therefore:

* To investigate which sexual side effects occur after EBRT and BT
* To investigate how many patients are affected
* To investigate if there is a time dependency for the severity of the sexual side effects
* To investigate if there is a dose dependency for the severity of the sexual side effects
* To find predicting and associated factors for the discovered sexual side effects to help identifying patients at risk

Background:

As mentioned above, very few studies have investigated sexual side effects aside from ED in EBRT patients. O'Neil et al found that out of 110 EBRT patients 5.2% reported to have orgasm associated UI; while, 28.3% of the 279 RP patients queried reported the problem [7]. Penile shortening have has consistently been found after RP [8]. However, after both brachytherapy and ERBT in conjunction with androgen deprivation therapy penile shortening have has also been described [9] . Sullivan et al. investigated ejaculatory profiles en men undergoing radiation therapy (RT), either EBRT, brachytherapy, or a combination of both [10]. They found that 5 years after RT 89% of the patients reported anejaculation. During the 5 years of follow up patients reported increasingly bad scores, as measured by the orgasm domain of the international index of erectile function (IIEF).

Research plan, participants, and methods:

Because of the apparent shortage of studies with the main aim of investigating sexual side effects other than ED after EBRT and BT, the investigators want conduct a single center cross-sectional questionnaire based study which will be comparable to our study on RP side effects [6]. The investigators hope to document how many patients are affected by UI during sexual stimulation, altered perception of orgasm, anejaculation, orgasm-associated pain, penile shortening, altered penile curvature, and penile sensory changes. Furthermore we want to identify predicting and associated factors to better understand why and when these side effects occur.

The study will start in September 2014 and the investigators anticipate to have completed data collection in December 2014. Initially the investigators plan to invite 20 patients to participate in interview sessions where they will be given the opportunity to contribute to the design of the questionnaire. When the final questionnaire is ready all suited patients will receive the questionnaire by mail. Initial non-responders will receive another questionnaire 4-6 weeks later in order to get as many answers as possible. In order to grant us permission to search the patients´ journals for background information all patients will receive an informed consent formula to sign.

Recruiting of patient and informed consent:

Patients will be identified through hospital records. Initially 10 EBRT patients and 10 BT patients will be contacted by telephone in order to arrange the interview sessions. The remaining patients will only be contacted by mail as described above. Patients will be informed of the purpose of the study and that the final publication of study result will be kept anonymous. Patients will be asked to state that they accept the publication.

The initial questionnaires will be accompanied by a letter explaining the importance of participating. One month after the questionnaires are expected to have been received by the patients a reminder will be send to non-responders.

Publication of results:

The final results will be published in a peer reviewed international journal as soon as possible. Should that not be possible the results will be made public on our hospitals internet homepage. Prevalence rates will be the main outcomes; while Univariate and multivariate logistic regression analyses will be used for the purpose of identifying associated and predicting factors.

Ethics:

The study will be carried out according to the rules stated in the declaration of Helsinki and Danish law concerning health care research. The study is approved by the Danish data protection agency and registered at clinicaltrials.org.

Hopefully this study can help adding valuable knowledge to an area that is largely undiscovered. In addition, the investigators expect these results to help draw a clearer picture of the pros and cons of RP, BT, and EBRT as treatments for localized prostate cancer. Finally, this study should help patients suffering sexual side effects after EBRT by making practitioners aware of their existence and providing them with knowledge to better inform future patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have received EBRT or BT with curative intent for localized prostate cancer.
* Only patients who have received EBRT or BT between 3 months and 5 years prior the start of the study will be enrolled.

Exclusion Criteria:

* Patients who had symptoms corresponding to the abovementioned side effects before EBRT

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients have received either external beam radiation therapy or brachie therapy as definitive treatment for localized prostate cancer between at Herlev hospital, Copenhagen, Denmark between 3 months and 5 years prior to being invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence during sexual activity | between 3 months to 5 years after intervention
  prevalence rate
penis shortening | between 3 months to 5 years after intervention
  prevalence rate
Orgasmic dysfunction | between 3 months to 5 years after intervention
  prevalence rate
anejaculation | between 3 months to 5 years after intervention
  prevalence rate
sensory changes in the penis | between 3 months to 5 years after intervention
  prevalence rate

SECONDARY OUTCOMES:
erectile functioning | between 3 months to 5 years after intervention
  intenational index of erectile function score
Urinary incontinence | between 3 months to 5 years after intervention
  international consultation of incontinence questionnaire
comorbidities | between 3 months to 5 years after intervention
  charlston comorbidity index
gastro intestinal side effects | between 3 months to 5 years after intervention
  prevalence rate

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sønksen, Professor, Study Chair — The unit for urological research, Herlev Hospital

REFERENCES:
- [Background] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013. Eur Urol. 2014 Jan;65(1):124-37. doi: 10.1016/j.eururo.2013.09.046. Epub 2013 Oct 6. PMID 24207135
- [Background] Tal R, Alphs HH, Krebs P, Nelson CJ, Mulhall JP. Erectile function recovery rate after radical prostatectomy: a meta-analysis. J Sex Med. 2009 Sep;6(9):2538-46. doi: 10.1111/j.1743-6109.2009.01351.x. Epub 2009 Jun 9. PMID 19515209
- [Background] Ficarra V, Novara G, Rosen RC, Artibani W, Carroll PR, Costello A, Menon M, Montorsi F, Patel VR, Stolzenburg JU, Van der Poel H, Wilson TG, Zattoni F, Mottrie A. Systematic review and meta-analysis of studies reporting urinary continence recovery after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):405-17. doi: 10.1016/j.eururo.2012.05.045. Epub 2012 Jun 1. PMID 22749852
- [Background] Robinson JW, Moritz S, Fung T. Meta-analysis of rates of erectile function after treatment of localized prostate carcinoma. Int J Radiat Oncol Biol Phys. 2002 Nov 15;54(4):1063-8. doi: 10.1016/s0360-3016(02)03030-4. PMID 12419432
- [Background] Ataman F, Zurlo A, Artignan X, van Tienhoven G, Blank LE, Warde P, Dubois JB, Jeanneret W, Keuppens F, Bernier J, Kuten A, Collette L, Pierart M, Bolla M. Late toxicity following conventional radiotherapy for prostate cancer: analysis of the EORTC trial 22863. Eur J Cancer. 2004 Jul;40(11):1674-81. doi: 10.1016/j.ejca.2003.12.027. PMID 15251156
- [Background] O'Neil BB, Presson A, Gannon J, Stephenson RA, Lowrance W, Dechet CB, Tward JD, Myers JB, Brant WO. Climacturia after definitive treatment of prostate cancer. J Urol. 2014 Jan;191(1):159-63. doi: 10.1016/j.juro.2013.06.122. Epub 2013 Sep 16. PMID 24050893
- [Background] Frey A, Sonksen J, Jakobsen H, Fode M. Prevalence and predicting factors for commonly neglected sexual side effects to radical prostatectomies: results from a cross-sectional questionnaire-based study. J Sex Med. 2014 Sep;11(9):2318-26. doi: 10.1111/jsm.12624. Epub 2014 Jul 4. PMID 24995845
- [Background] Frey AU, Sonksen J, Fode M. Neglected side effects after radical prostatectomy: a systematic review. J Sex Med. 2014 Feb;11(2):374-85. doi: 10.1111/jsm.12403. Epub 2013 Nov 25. PMID 24267516
- [Background] Eylert MF, Bahl A, Persad R. Do we need to obtain consent for penile shortening as a complication of treatment for organ-confined prostate cancer? BJU Int. 2012 Nov;110(10):1491-500. doi: 10.1111/j.1464-410X.2012.11102.x. Epub 2012 Apr 23. PMID 22520266
- [Background] Sullivan JF, Stember DS, Deveci S, Akin-Olugbade Y, Mulhall JP. Ejaculation profiles of men following radiation therapy for prostate cancer. J Sex Med. 2013 May;10(5):1410-6. doi: 10.1111/jsm.12101. Epub 2013 Feb 22. PMID 23433425